CLINICAL TRIAL: NCT00440960
Title: Anesthesia in Flexible Bronchoscopy for Lung Cancer Diagnostic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Pompeia (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 0002.0.297.000-06
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Lung Cancer
Keywords: alfentanil; anesthesia; bronchoscopy; lidocaine; midazolam; propofol.
MeSH Terms: conditions — Lung Neoplasms | interventions — Propofol; Midazolam; Alfentanil; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: propofol
Drug: midazolam
Drug: alfentanil
Drug: lidocaine

SUMMARY:
The objective of the study was to establish which anesthetic procedure used during flexible bronchoscopy has the lowest index of complications.

DETAILED DESCRIPTION:
This prospective randomized study analyzed 80 patients that underwent flexible bronchoscopy. Patients were randomly assigned to four groups of 20 patients each according to the anesthetic combination used: 200 mg topical lidocaine (LID group); 200 mg topical lidocaine and 2 mg/kg propofol (PPF group); 200 mg topical lidocaine and 20 mcg/kg alfentanil (ALF group); or 200 mg topical lidocaine and 0.05 mg/kg midazolam (MID group). Scores were assigned to patients according to the different variables observed during the endoscopic procedure; the lower the score, the lower the complication index.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study were referred to FBC for the investigation of bronchial carcinoma (diagnostic procedure).
* Patients included in the study were classified as ASA I, II and II according to the anesthetic risk classification of the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* ASA IV classification of anesthesiology risk
* procedure that lasted longer than 15 minutes
* indication of therapeutic bronchoscopy
* cardiac arrhythmia and / or hypoxemia detected at admission.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andre GS Leite, PhD, Principal Investigator — Brazilian Society of Thoracic Surgery
Locations (3):
- Brazil (3):
  - Hospital Pompeia, Caxias do Sul, Rio Grande do Sul
  - Hospital Medianeira, Caxias do Sul, Rio Grande do Sul
  - General Hospital of Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul

REFERENCES:
- [Background] Pue CA, Pacht ER. Complications of fiberoptic bronchoscopy at a university hospital. Chest. 1995 Feb;107(2):430-2. doi: 10.1378/chest.107.2.430. PMID 7842773
- [Result] Barr J, Egan TD, Sandoval NF, Zomorodi K, Cohane C, Gambus PL, Shafer SL. Propofol dosing regimens for ICU sedation based upon an integrated pharmacokinetic-pharmacodynamic model. Anesthesiology. 2001 Aug;95(2):324-33. doi: 10.1097/00000542-200108000-00011. PMID 11506101
- [Result] Schaeuble J, Heidegger T, Gerig HJ, Ulrich B, Schnider TW. Comparision of etomidate and propofol for fibreoptic intubation as part of an airway management algorithm:a prospective, randomizes, double-blind study. Eur J Anaesthesiol. 2005 Oct;22(10):762-7. doi: 10.1017/s0265021505001262. PMID 16211735
- [Result] Amitai Y, Zylber-Katz E, Avital A, Zangen D, Noviski N. Serum lidocaine concentrations in children during bronchoscopy with topical anesthesia. Chest. 1990 Dec;98(6):1370-3. doi: 10.1378/chest.98.6.1370. PMID 2245677
- [Result] Koyama S, Koh H, Noda K, Tagami N, Asada A. [A comparison of the incidence of postoperative nausea and vomiting after propofol-fentanyl anesthesia and that after nitrous oxide-isoflurane anesthesia]. Masui. 1998 Mar;47(3):286-9. Japanese. PMID 9560538
- [Result] Hautmann H, Bauer M, Pfeifer KJ, Huber RM. Flexible bronchoscopy: a safe method for metal stent implantation in bronchial disease. Ann Thorac Surg. 2000 Feb;69(2):398-401. doi: 10.1016/s0003-4975(99)01398-3. PMID 10735670
- [Result] Cartwright CR, Henson LC, Ward DS. Effects of alfentanil on the ventilatory response to sustained hypoxia. Anesthesiology. 1998 Sep;89(3):612-9. doi: 10.1097/00000542-199809000-00009. PMID 9743396
- [Result] Pereira W Jr, Kovnat DM, Snider GL. A prospective cooperative study of complications following flexible fiberoptic bronchoscopy. Chest. 1978 Jun;73(6):813-6. doi: 10.1378/chest.73.6.813. PMID 657853
- [Result] Clarkson K, Power CK, O'Connell F, Pathmakanthan S, Burke CM. A comparative evaluation of propofol and midazolam as sedative agents in fiberoptic bronchoscopy. Chest. 1993 Oct;104(4):1029-31. doi: 10.1378/chest.104.4.1029. PMID 8404160